CLINICAL TRIAL: NCT00964496
Title: Long-term Effects of Thalidomide for Recurrent Gastrointestinal Bleeding Due to Vascular Malformation : An Open-label, Randomized, Parallel Controlled Study
Brief Title: Long-term Effects of Thalidomide for Recurrent Gastrointestinal Bleeding Due to Vascular Malformation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Zhizheng Ge, MD. Ph.D ,Professor ,Shanghai Ren Ji Hospital, Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjyyxhk3015
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2009-08

CONDITIONS: Obscure Gastrointestinal Bleeding; Angiodysplasia; Gastric Antral Vascular Ectasia; Thalidomide
Keywords: vascular malformation; gastrointestinal bleeding; thalidomide
MeSH Terms: conditions — Angiodysplasia; Gastric Antral Vascular Ectasia; Vascular Malformations; Gastrointestinal Hemorrhage | interventions — Thalidomide; Iron; ferrous succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thalidomide Group (Active Comparator)
  Interventions: Drug: Thalidomide
- Iron-controlled Group (Other)
  Interventions: Drug: Iron

INTERVENTIONS:
Drug: Thalidomide — Patients were randomly assigned to receive a four-month course of 25 mg of thalidomide (Pharmaceutical Co., Ltd. of Chang-zhou, China). Medications were taken orally four times daily at 6 a.m., 12 noon, 6 p.m., and 10 p.m.
  Other Names: Softenon;
  Arms: Thalidomide Group
Drug: Iron — Patients were randomly assigned to receive a four-month course of 100 mg of iron (Pharmaceutical Co., Ltd. of Nanjing, China). Medications were taken orally four times daily at 6 a.m., 12 noon, 6 p.m., and 10 p.m.
  Other Names: Ferrous Succinate Tablets
  Arms: Iron-controlled Group

SUMMARY:
Background: Repeated episodes of bleeding from gastrointestinal vascular malformations refractory to endoscopic or surgical therapy often pose a major therapeutic challenge.

Methods: The investigators performed a randomized, parallel controlled study of thalidomide as a therapy for recurrent gastrointestinal bleeding due to vascular malformation. Patients with at least six episodes of bleeding in the prior year due to vascular malformation were randomly grouped, prescribed a four-month regimen of either 25 mg of thalidomide or 100 mg of iron orally four times daily, and monitored for at least one year. The primary end point was defined as the patients whose rebleeds decreased from baseline by ≥ 50% at 12 months and the cessation of bleeding. Rebleeding was defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment. Secondary outcomes included the participants dependent on blood transfusions and changes from baseline in transfused packed red cell units, bleeding episodes, bleeding durations, and hemoglobin levels at 12 months. Statistical significance was defined at P < 0.05.

DETAILED DESCRIPTION:
Protocol Description:

This is an exploratory, randomized, parallel controlled study of thalidomide for recurrent gastrointestinal bleeding from vascular malformations. Informed consent was taken from all subjects and the Institute Ethics Committee approved the study protocol. All procedures were in accordance with the Declaration of Helsinki. The study was supported by no pharmaceutical funding.

Study design and Intervention:

From Nov. 2004 to Nov. 2007, patients with repeated episodes of chronic gastro-intestinal bleeding due to vascular malformations identified by oesophagogastroduodenoscopy, capsule endoscope or double-balloon endoscope were enrolled (according our enrollment criteria).

The patients were randomly assigned to receive a four-month course of either 25 mg of thalidomide or 100mg iron orally at daily time 6 a.m.,12 noon,6 p.m. and 10 p.m., respectively.

Randomization was performed through the proc plan procedure of Statistical Analysis Software (SAS), using the method of randomly permuted blocks of 4. Within each block, the number of patients allocated to each of the two treatments was equal. Each patient who met the inclusion criteria was consecutively assigned a random number in chronological order, which allocated him or her to one of the treatment groups. A blinded research nurse supervised patient randomization and drug administration.

In the case of an adverse event, the study medication was temporarily or permanently discontinued based on subject inclination and toxicity intolerance. Concomitant therapies, such as blood transfusions and other symptomatic treatments like iron supplementation, were performed in both groups as necessary during the four-month treatment and subsequent follow-up periods. Blood transfusion was indicated and recorded when the hemoglobin (Hb) level reached < 7.0 g/dl. Red-cell transfusions were administered according to patient Hb level as follows: 2 units were administered for 6.1 g/dl ≥ Hb ≤ 7.0 g/dl, 3 units for 5.1 g/dl ≥ Hb ≤ 6.0 g/dl, and 4 units for Hb < 5.0 g/dl. Iron was provided for patients with 7.0 g/dl ≥ Hb ≤ 11.0 g/dl. After the four-month treatment course, all patients discontinued study medications except for cases where symptomatic treatments were necessary as described above.

Assessment of response and adverse events:

The primary end point was defined as the patients whose rebleeds decreased from baseline by ≥ 50% at 12 months and the cessation of bleeding. Rebleeding was defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment. Secondary outcomes included the participants dependent on blood transfusions and changes from baseline in transfused packed red cell units, bleeding episodes, bleeding durations, and hemoglobin levels at 12 months.

Adverse events included any unfavorable change in health, including abnormal laboratory findings, during the study or follow-up period.

Evaluation of Patients and Follow-up:

* Certified research nurses collected information on the demographics and medical and social histories of all patients enrolled in the study.
* After screening and baseline evaluations, the patients were closely monitored in the hospital for at least one week. They were then followed twice monthly during the four-mouth course of treatment and once a month thereafter.
* Clinical follow-up was performed by qualified doctors. At all visits, the bleeding-related parameters (number and duration), a physical examination was performed and laboratory values were obtained for FOBT, complete blood counts, serum chemistries, and hepatic and renal function. Neuropathy and other adverse events were also assessed.
* Patients were advised to refrain from any other non-prescribed medicines, especially rebleeding-related medications such as aspirin, nonsteroidal antiinflammatory drugs (NSAIDs), anti-platelet drugs, anticoagulants, and Chinese medications (with salicylates), gingko, or Echinacea.

Measurement of Vascular Endothelial Growth Factor (VEGF) in Sera:

Laboratory assays for VEGF were performed at baseline and after the four-month treatment course in the thalidomide group, by a technician blinded to the assignment and final assessment. Three milliliters of serum of peripheral venous blood samples were centrifuged (3000 r/min at 4°C, 10 min), extracted, separated into freezing tubes, and stored at -70°C for no more than 4 months. Plasma VEGF levels (in pg/ml) were determined in duplicate using sandwich ELISA kits (R&D Systems, USA) in a laboratory of the Shanghai Research Institute of Digestive Disease. Samples from each patient were batch-tested in a single run. For quality control, all samples were retested two more times in a subsequent run to confirm the results of the first run.

Statistical Analysis:

To our knowledge, no similar such study has previously been performed, and we were thus unable to refer to published studies to determine our samples. To this end, we performed an unpublished preliminary study. Response in the iron-control group and thalidomide group reached 10% and 80%, due to loose inclusion criteria (bleeding history was not restricted). For this study, we estimated that the primary outcome (the proportion of subjects whose number of yearly bleeds had decreased by ≥ 50%) would occur in 10% of the control group and 80% of the thalidomide group patients. An equally divided sample of 11 subjects was deemed sufficient for detecting the primary end point, with a type I error (two-sided) of 5% and a power of 90%. Assuming a 10% volunteer attrition rate to follow-up, we established a target sample size of 13 per group (calculated with nquery advisor software 5.0).

Analyses of the responses and adverse events were performed on all registered patients according to the intention-to-treat principle. Statistical analysis was performed by a blinded biostatistician with the Statistical Product and Service Solutions (SPSS) 13.0 software package. We simultaneously analyzed the primary endpoint of the full analysis set (FAS) and per protocol set (PPS). Continuous variables were compared using a two-sample independent t-test or Wilcoxon rank-sum test. Categorical variables were compared using the chi-squared and Fisher's exact tests. A paired t-test was employed to compare differences in plasma VEGF levels before and after thalidomide treatment. The Breslow-Day test was used to test for the heterogeneity of treatment effects across strata. All reported P-values are two-sided. Data are reported as the mean ± standard deviation (SD) or median (range) for continuous variables and number (%) for categorical variables. Since adjustments to the control group were minimal, we also reported point estimates and 95% confidence intervals (CIs). For all outcomes, a P-value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-85 years; women were post-menopausal, post-tubal ligation, or on some form of birth control like long-term laying up contraceptive ring or using condom;
* History of at least six documented gastrointestinal bleeding episodes in the year prior to randomization, which were refractory or inaccessible to endoscopic therapy or surgical ectomy;
* Confirmed diagnosis of vascular malformation by esophagogastroduodenoscopy (EGD), capsule endoscope (CE), double-balloon endoscope (DBE), or colonoscopy, but no obvious infectious, neoplastic, or other specific diagnosis;
* Angiodysplasia at endoscopy characterized by focal or diffused venous/capillary lesions presenting as bright red ectatic vessels or pulsatile red protrusions, with surrounding venous dilatation or patchy erythema with or without oozing;
* Endoscopic appearance of GAVE (also known as watermelon stomach), indicated by longitudinal antral folds converging on the pylorus, containing visible columns of tortuous red ecstatic vessels.

Exclusion Criteria:

* Patients were excluded if their bleeding history were less than 1 year;
* if they had cirrhotic or portal hypertension gastropathy; severe co-morbidities of cardiac, pulmonary, renal, liver, hematological, rheumatologic disorders, or uncontrollable diabetes mellitus or hypertension;
* if they had a history of severe bilateral peripheral neuropathy or seizure activity, thromboembolic disease, known thalidomide or iron allergy, or prior treatment of gastrointestinal bleeding with thalidomide;
* if they had a history of treatment with any dose of systemic or oral topical corticosteroids or aspirin, NSAIDs, anti-platelet drugs, anticoagulants, or Chinese medications (with salicylates), gingko, or Echinacea, or other putative immunomodulators or anti-angiogenic agents;
* Currently pregnant or lactating or currently undergoing systemic cancer chemotherapy or receiving radiation
* if they were undergoing systemic cancer chemotherapy or receiving radiation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-11; Primary Completion 2007-11 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhizheng Ge, MD. Ph.D, Principal Investigator — Shanghai Ren Ji Hospital

REFERENCES:
- [Background] Jacobson JM, Greenspan JS, Spritzler J, Ketter N, Fahey JL, Jackson JB, Fox L, Chernoff M, Wu AW, MacPhail LA, Vasquez GJ, Wohl DA. Thalidomide for the treatment of oral aphthous ulcers in patients with human immunodeficiency virus infection. National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group. N Engl J Med. 1997 May 22;336(21):1487-93. doi: 10.1056/NEJM199705223362103. PMID 9154767
- [Background] Bauditz J, Schachschal G, Wedel S, Lochs H. Thalidomide for treatment of severe intestinal bleeding. Gut. 2004 Apr;53(4):609-12. doi: 10.1136/gut.2003.029710. PMID 15016759
- [Background] Shurafa M, Kamboj G. Thalidomide for the treatment of bleeding angiodysplasias. Am J Gastroenterol. 2003 Jan;98(1):221-2. doi: 10.1111/j.1572-0241.2003.07201.x. No abstract available. PMID 12526972
- See also: Approved drug page at FDA's Drugs@FDA web site. — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Overview&DrugName=THALOMID&CFID=21312735&CFTOKEN=394df9d228870faa-4F4FD0A6-1372-5AE1-6AD225831B3F092E

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From November 2004 to November 2007, a total of 59 subjects were assessed for eligibility at Shanghai Ren Ji Hospital, China.
Pre-assignment Details: Among the 59 patients, two refused to enter the protocol and two other were excluded owing to severe associated disease with short life expectancy. Therefore, 55 patients were enrolled in our study.
Groups:
- Thalidomide Group: interventions administered (dosage, 100mg; dosage form, 25mg; frequency of administration, 4 times daily at 6 a.m., 12 noon, 6 p.m., and 10 p.m)
- Iron-controlled Group: interventions administered (dosage, 400mg; dosage form, 100mg; frequency of administration, 4 times daily at 6 a.m., 12 noon, 6 p.m., and 10 p.m)
Period: Overall Study
Arm/Group | Thalidomide Group | Iron-controlled Group
Started | 28 | 27
Completed | 26 | 26
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thalidomide Group | Iron-controlled Group | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  China | 28 | 27 | 55
Location [Number; unit: participants]
  Multiple | 13 | 14 | 27
  Single | 15 | 13 | 28
Outcome [Number; unit: participants]
  Completion of study | 26 | 26 | 52
  Incomplete study | 2 | 1 | 3
Transfusion dependence [Number; unit: participants]
  dependent | 14 | 14 | 28
  independent | 14 | 13 | 27
Ways of diagnose [Number; unit: participants]
  Capsule endoscopy | 24 | 24 | 48
  Enteroscopies | 2 | 2 | 4
  Gastroscopy | 2 | 1 | 3
Activated partial thromboplastin time (APTT) [Mean (Standard Deviation); unit: seconds] | 27.4929 (6.4430) | 28.0667 (5.9947) | 27.7745 (6.1760)
Follow-up time [Mean (Standard Deviation); unit: months] | 34.9286 (13.73810) | 36.1481 (13.49274) | 35.5273 (13.50563)
Glutamic-pyruvic transaminase (GPT) [Mean (Standard Deviation); unit: IU/L] | 24.8143 (13.4963) | 25.2019 (14.1123) | 25.0045 (12.4753)
History of bleeding time [Median (Full Range); unit: years] | 5 (4.1404) [1 to 21] | 3 (4.4331) [1 to 20] | 5 (4.2552) [1 to 21]
Mean corpuscular volume (MCV) [Mean (Standard Deviation); unit: femtoliter] | 76.8000 (3.9711) | 75.2444 (4.4130) | 76.0364 (4.2282)
Mean Corpuscular Hemoglobin Concentration [Mean (Standard Deviation); unit: g/L] | 295.8571 (15.2624) | 299.0000 (13.3012) | 297.4000 (14.2888)
Platelet count (PLT) [Mean (Standard Deviation); unit: 10^9/L] | 206.4536 (53.1686) | 197.7111 (60.0851) | 202.1618 (56.3131)
Pre- packed red cell units transfused per year [Mean (Standard Deviation); unit: milliliter] — Total packed red cell units transfused per year(milliliter) before randomization in transfusion dependent subjects.
  milliliter | 1928.57 (763.02) | 1985.71 (766.47) | 1957.14 (751.01)
Pre-bleeding duration [Mean (Standard Deviation); unit: days] | 8.8214 (3.0799) [5 to 20] | 8.7407 (4.5029) [3 to 21] | 8.7818 (3.8088) [3 to 21]
Pre-treatment hemoglobin level [Mean (Standard Deviation); unit: g/dl] | 6.4000 (1.7904) | 5.9919 (1.5304) | 6.1996 (1.6652)
Prothrombin time-international normalized ratio (PT-INR) [Mean (Standard Deviation); unit: seconds] | 1.0550 (0.1530) | 1.0989 (0.1533) | 1.0765 (0.1534)
Serum creatinine [Mean (Standard Deviation); unit: mg/dl] | 77.5536 (20.9532) | 88.9296 (24.2665) | 83.1382 (23.1514)
Total bilirubin [Mean (Standard Deviation); unit: μmol/L] | 9.1607 (4.4212) | 9.1407 (4.1196) | 9.1509 (4.2361)
White blood cell (WBC) [Mean (Standard Deviation); unit: 10^9/L] | 6.4429 (1.5704) | 6.5926 (1.7389) | 6.5164 (1.6416)
pre-bleeding episodes per year [Mean (Standard Deviation); unit: bleeding episodes] | 13.96 (3.383) [7 to 19] | 13.96 (3.469) [7 to 21] | 13.96 (3.394) [7 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Participants Whose Rebleeds Decreased From Baseline by ≥ 50% at 12 Months
Description: The primary end point was defined as the patients whose rebleeds decreased from baseline by ≥ 50% at 12 months. Reduction of rebleeds = [(total bleeding episode at 12 months - total bleeding episodes at a year before randomization)/total bleeding episodes at a year before randomization(baseline)]*100%. Rebleeding was defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment.
Time Frame: baseline and 12 months
Measure: Number; unit: participants
Arm/Group | Thalidomide Group | Iron-controlled Group
Number analyzed (Participants) | 28 | 27
participants | 20 | 1
Statistical Analysis 1: Comparison: Thalidomide Group vs Iron-controlled Group; Null hypothesis (H0): Thalidomide 100 mg per day is equivalence to iron 400 mg per day with regard to the participants whose rebleeds decreased from baseline by ≥ 50% at 12 months. Alternative hypothesis (Ha): Thalidomide 100 mg per day is non-equivalent to iron 400 mg per day with regard to the participants whose rebleeds decreased from baseline by ≥ 50% at 12 months. Comparisons were performed with the use of the chi-square test, Fisher's exact test; Test type: Superiority or Other; p = 0.00000013, Fisher Exact — P<0.05 was considered as statistical different, while P>0.05 was considered as no statistical significance between two groups. All reported P values are two-sided; Differences in proportions = 0.677, 95% CI 2-sided [0.547 to 0.807]

2. Secondary Outcome: Change From Baseline in Hemoglobin (Hb) Level at 12 Months
Description: The change from baseline in average hemoglobin (Hb) level(tested every month) at 12 months.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Thalidomide Group | Iron-controlled Group
Number analyzed (Participants) | 28 | 27
g/L | 3.06 (2.08) | -0.01 (1.32)
Statistical Analysis 1: Comparison: Thalidomide Group vs Iron-controlled Group; Null hypothesis (H0): Thalidomide 100 mg per day is equivalence to iron 400 mg per day with regard to the change from baseline in hemoglobin level at 12 months. Alternative hypothesis (Ha): Thalidomide 100 mg per day is non-equivalent to iron 400 mg per day with regard to the change from baseline in hemoglobin level at 12 months. Comparisons were performed with the use of the independent-samples t test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.08, 95% CI 2-sided [-4.02 to -2.13]

3. Secondary Outcome: Change From Baseline in Bleeding Episodes at 12 Months
Description: The Change from baseline in bleeding episodes at 12 months
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: bleeding episodes
Arm/Group | Thalidomide Group | Iron-controlled Group
Number analyzed (Participants) | 28 | 27
bleeding episodes | -9.36 (4.31) | 1.41 (2.74)
Statistical Analysis 1: Comparison: Thalidomide Group vs Iron-controlled Group; Null hypothesis (H0): Thalidomide 100 mg per day is equivalence to iron 400 mg per day with regard to the change from baseline in bleeding episodes at 12 months. Alternative hypothesis (Ha): Thalidomide 100 mg per day is non-equivalent to iron 400 mg per day with regard to the change from baseline in bleeding episodes at 12 months. Comparisons were performed with the use of the independent-samples t test; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.95, 95% CI 2-sided [6.00 to 9.90]

4. Secondary Outcome: Change From Baseline in Bleeding Duration at 12 Months
Description: The change from baseline in bleeding duration at 12 months
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thalidomide Group | Iron-controlled Group
Number analyzed (Participants) | 28 | 27
days | 5.2 (3.0) | 0.8 (5.1)
Statistical Analysis 1: Comparison: Thalidomide Group vs Iron-controlled Group; Null hypothesis (H0): Thalidomide 100 mg per day is equivalence to iron 400 mg per day with regard to the change from baseline in bleeding duration at 12 months. Alternative hypothesis (Ha): Thalidomide 100 mg per day is non-equivalent to iron 400 mg per day with regard to the change from baseline in bleeding duration at 12 months. Comparisons were performed with the use of the independent-samples t test; Test type: Superiority or Other; p = 0.00024740, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.40, 95% CI 2-sided [2.15 to 6.64]

5. Secondary Outcome: Participants Dependent on Blood Transfusions
Description: Numbers of participants dependent on blood transfusions
Time Frame: 52 months
Population: 55 patients were enrolled in our study. One in iron-controlled group refused to continue for personal reason after 8 months, two other in thalidomide plus iron group refused to take study medications after 4 weeks treatment due to leukopenia and unexplained somnolence. Analysis was performed according to Intention-to-Treat principle.
Measure: Number; unit: participants
Arm/Group | Thalidomide Group | Iron-controlled Group
Number analyzed (Participants) | 28 | 27
participants | 3 | 13
Statistical Analysis 1: Comparison: Thalidomide Group vs Iron-controlled Group; Null hypothesis (H0): Thalidomide 100 mg per day is equivalence to iron 400 mg per day with regard to the participants dependent on blood transfusions. Alternative hypothesis (Ha): Thalidomide 100 mg per day is non-equivalent to iron 400 mg per day with regard to the participants dependent on blood transfusions. Comparisons were performed with the use of the chi-square test, Fisher's exact test; Test type: Superiority or Other; p = 0.00298881, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Differences in proportions = -0.374, 95% CI 2-sided [-0.563 to -0.185]

6. Secondary Outcome: Change From Baseline in Total Transfused Red Cell Requirements at 12 Months
Description: Change of total transfused red cell requirements at 12 months after randomization from one year before baseline in transfusion dependent patients
Time Frame: baseline and 12 months
Population: There are 14 participants depended on blood transfusion in each group
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Thalidomide Group | Iron-controlled Group
Number analyzed (Participants) | 14 | 14
milliliter | -1585.71 (446.97) | -28.57 (106.90)
Statistical Analysis 1: Comparison: Thalidomide Group vs Iron-controlled Group; Null hypothesis (H0): Thalidomide 100 mg per day is equivalence to iron 400 mg per day with regard to the change from baseline in total transfused red cell requirements at 12 months. Alternative hypothesis (Ha): Thalidomide 100 mg per day is non-equivalent to iron 400 mg per day with regard to the change from baseline in total transfused red cell requirements at 12 months. Comparisons were performed with the use of the independent-samples t test; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1557.14, 95% CI 2-sided [1294.53 to 1819.76]

7. Primary Outcome: Cessation of Bleeding
Description: The cessation of bleeding was defined as repeated negative faecal occult blood test (FOBT) (monoclonal colloidal gold color technology) during our observation period. Rebleeding was defined based on a positive FOBT at any visit after treatment.
Time Frame: 52 months
Measure: Number; unit: participants
Arm/Group | Thalidomide Group | Iron-controlled Group
Number analyzed (Participants) | 28 | 27
participants | 13 | 0
Statistical Analysis 1: Comparison: Thalidomide Group vs Iron-controlled Group; Null hypothesis (H0): Thalidomide 100 mg per day is equivalence to iron 400 mg per day with regard to the cessation of bleeding. Alternative hypothesis (Ha): Thalidomide 100 mg per day is non-equivalent to iron 400 mg per day with regard to the cessation of bleeding. Comparisons were performed with the use of the chi-square test, Fisher's exact test; Test type: Superiority or Other; p = 0.00003962, Fisher Exact; Differences in proportions = 0.464, 95% CI 2-sided [0.28 to 0.649]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during 4-month treatment and thereafter medium 39 months (range: 8 to 52 months) of follow-up.
Description: Adverse events were considered if any uncomfortable symptoms occur and relevant to our study medications. Severe adverse events (SAE's) were considered if the complained symptoms resulted in more hospitalization or that threaten the patients lives.
Arm/Group | Thalidomide Group | Iron-controlled Group
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 20/28 | 9/27
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide Group (N=28) | Iron-controlled Group (N=27)
Abdominal distension (Gastrointestinal disorders) | 1 (9) | 1 (12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (7)
Bitter taste (Gastrointestinal disorders) | 2 (10) | 0 (0)
Blurred vision (Eye disorders) | 1 (5) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (92) | 3 (18)
Dizziness (General disorders) | 6 (82) | 2 (10)
Dryness of eye (Eye disorders) | 1 (5) | 0 (0)
Fatigue (General disorders) | 9 (72) | 3 (12)
Hands tremble (Nervous system disorders) | 1 (4) | 0 (0)
Headache (Nervous system disorders) | 1 (8) | 0 (0)
Increase in vaginal discharge (Endocrine disorders) | 1 (60) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Nuasea (Gastrointestinal disorders) | 0 (0) | 1 (5)
Numb limb (Nervous system disorders) | 1 (6) | 0 (0)
Otalgia (Ear and labyrinth disorders) | 1 (5) | 0 (0)
Peripheral edema (Vascular disorders) | 4 (16) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shingles zoster Infection (Infections and infestations) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (8) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 3 (18)
Thrombopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (4)

LIMITATIONS AND CAVEATS:
Single center, open-label study; lack of placebo pills, make it impossible on equality of dosages between two groups; lack of dose response assessment either in patients or assays of serum vascular endothelial growth factor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes